CLINICAL TRIAL: NCT03575494
Title: Oral Health Status and Unexplained Female Infertility
Brief Title: Relationship Between Oral Health Status and Unexplained Female Infertility in Turkish Population
Status: Withdrawn | Type: Observational
Why Stopped: this study does not need to get a clinicaltrials number
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Recep Tayyip Erdogan University Faculty of Dentistry, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 40465587-177
Record Dates: First submitted 2018-06-22; First posted 2018-07-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Dental Caries; Female Infertility
MeSH Terms: conditions — Dental Caries; Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- female infertility: Women who had regular menses and can't conceive despite a long-term regular sexual intercourse for more than 12 months
  Interventions: Other: Intraoral and Radiographic Dental Examination
- healthy: healthy patients who had minimum two normal pregnancies
  Interventions: Other: Intraoral and Radiographic Dental Examination

INTERVENTIONS:
Other: Intraoral and Radiographic Dental Examination — (ORTHOPANTOMOGRAPH® OP300 PANORAMIC, Instrumentarium Dental, Tuusula, Finland,63 kVp, 0.8 mA, 0.5 s).

SUMMARY:
Periodontal diseases and dental caries are initiated by a pathogenic biofilm, in a susceptible host, affecting the tooth periodontium and hard tissues. Its possible association with many biologic systems has been studied. In this study, researchers investigated association between oral health and female infertility, and what is the biological rationale for such relationship.

DETAILED DESCRIPTION:
Power analysis was performed with the G-Power software package to determine sample size.

To cover possible data loss, 10% of a group were added to each group. Medical and dental examination will be performed both of control and experimental groups. In dental examination decayed, missing, or filled teeth (DMFT) index will be used according to World Health Organization (WHO 1997) criteria. All teeth were visually using the International Caries Detection and Assessment System (ICDAS-II).

To analyze the correlation between oral health status and female infertility linear regression test and for comparison of both the groups (case and control), two sample t test and chi square test were used.

ELIGIBILITY:
Inclusion Criteria:

* Women who had regular menses and can't conceive despite a long-term regular sexual intercourse for more than 12 months
* Women with normal hormone values and uterine cavity with at least one healthy fallopian tube.
* All male partners have a semen specimen with minimum 5 million motile sperm in the ejaculate.
* The control group members have minimum two normal pregnancies

Exclusion Criteria:

* Patients who have history of f; hydrosalpinx, polycystic ovarian syndrome, endometriosis grade 3-4, thyroid disease, tubal surgery, hyperprolactinemia, autoimmune diseases, diabetes mellitus, uterine/cervical anomalies, active liver disease, cardiovascular disease, premature ovarian failure, smoking and alcohol consumption, poor socioeconomic level, HIV-infected, obesity (body mass index ≥ 30 kg/m2), chronic upper respiratory tract diseases and dental fluorosis.
* Patients using fluoride supplements and orthodontic appliances

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients were aged from 18 to 35 years, 100 females
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-04-15 (Estimated); Primary Completion 2019-04-15 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
female infertility | 12 months
  Women with normal hormone values and uterine cavity with at least one healthy fallopian tube.
  All male partners have a semen specimen with minimum 5 million motile sperm in the ejaculate.

SECONDARY OUTCOMES:
dental examination | 1 Day
  All teeth were visually using the International Caries Detection and Assessment System (ICDAS-II). The chosen sites were recorded as:
  0 = sound;
  1. = first visible sign of noncavitated lesion seen only when the tooth is dried;
  2. = visible noncavitated lesion seen when wet and dry;
  3. = microcavitation in enamel;
  4. = noncavitated lesion extending into dentine seen as an undermining shadow;
  5. = small cavitated lesion with visible dentine: less than 50% of surface;
  6. = large cavitated lesions with visible dentine in more than 50% of the surface. A single calibrated examiner measured probing depth-PD, clinical attachment level- CAL, plaque (Pl), and gingival indices (GI), bleeding on probing (BOP) at four sites per tooth using a manual periodontal probe (PCPUNC, Hu-Friedy, Chicago, IL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yıldız Telatar, Principal Investigator — Recep Tayyip Erdogan University Dentistry Faculty
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be available within 6 months of study finishing

REFERENCES:
- [Background] Khanna SS, Dhaimade PA, Malhotra S. Oral Health Status and Fertility Treatment Including IVF. J Obstet Gynaecol India. 2017 Dec;67(6):400-404. doi: 10.1007/s13224-017-1025-0. Epub 2017 Jun 20. PMID 29162952
- See also: Oral Health Status and Fertility Treatment — http://www.ncbi.nlm.nih.gov/pubmed/29162952